CLINICAL TRIAL: NCT03898518
Title: The Effects of a 12-week Jump Rope Exercise Program on Body Composition, Insulin Sensitivity, and Academic Self-efficacy in Obese Prehypertensive Adolescent Girls
Brief Title: The Effects of a Jump Rope Exercise Program on Body Composition and Self-efficacy in Obese Adolescent Girls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University (Other)
Collaborators: Chonnam National University (Other); University of Nebraska (Other)
Responsible Party: Principal Investigator, Won-mok son, Principal Investigator, Pusan National University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UNOVRLJRSE
Record Dates: First submitted 2019-03-29; First posted 2019-04-02 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Prehypertension; Blood Pressure; Abdominal Obesity; Self Efficacy; Adiposity; Insulin Sensitivity
Keywords: adolescence; exercise; body composition; insulin sensitivity; obesity; academic self-efficacy
MeSH Terms: conditions — Prehypertension; Obesity, Abdominal; Obesity; Insulin Resistance; Motor Activity

STUDY DESIGN:
Intervention Model Description: exercise intervention group, control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): The control group was in the facility for all jump rope exercise sessions but did not participate in the exercise intervention.
- Experimental Group (Experimental): The experimental group performed the jump rope exercise intervention.
  Interventions: Other: 12-week jump rope exercise program

INTERVENTIONS:
Other: 12-week jump rope exercise program — Each jump rope exercise session of the program was performed for 50 minute, with a 5 minute warm-up and cool-down. Sessions were performed once a day, 5 days a week, for 12 weeks. The program consisted of various main jump rope exercises (1 line 2 jump, jumping feet together, running jumping, open side jump, open back and forth jump, rock paper scissor jump). The warm-up and cool-down consisted of static stretching, walking, and jogging. Intensity of exercise was gradually increased form 40-50% heart rate reserve (HRR) in weeks 1-4 and 60-70% HRR in weeks 9-12. Each training session was supervised by the researchers. Ever subject wore a heart rate monitor during the whole training session in order to maintain the designated training intensity.
  Arms: Experimental Group

SUMMARY:
The purpose of this study was to examine the impact of a 12-week jump rope exercise program on body composition, blood pressure, insulin resistance, and academic self-efficacy in prehypertensive adolescent obese girls. Forty-eight prehypertensive adolescent obese girls participated in this study. The girls were randomly divided into the jump rope exercise intervention group (EX, n=24) and control group (CON, n=24). The EX group performed a jump rope training program at 40-70% of their heart rate reserve (HRR) 5 days/week for 12 weeks (sessions 50 minutes in duration). The CON group did not participate in any structure or unstructured exercise protocol. Blood pressure, body fat percentage, waist circumference, blood glucose and insulin, homeostatic model assessment - insulin resistance, and Academic Self-Efficacy were measured before and after the 12-weeks study.

ELIGIBILITY:
Inclusion Criteria:

* prehypertensive
* sedentary (no regular exercise training or physical activity within the last year)
* no weight loss diet during the last six months
* obese

Exclusion Criteria:

* pregnancy
* chronic disease
* daily medication use

Ages: 14 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2010-10-03 (Actual); Primary Completion 2011-02-23 (Actual); Study Completion 2011-12-06 (Actual)

PRIMARY OUTCOMES:
Body Fat | 12 weeks
  Body fat percentage was measured to the nearest 0.1%.
Blood Pressure | 12 weeks
  Blood pressure was measured in duplicate using an automated sphygmomanometer. The average of the was recorded as the resting blood pressure. Both systolic and diastolic blood pressure were recorded.
Body Mass | 12 weeks
  Body mass was measured to nearest 0.1kg.
Height | 12 weeks
  Height was measured to the nearest 1 cm.
Waist Circumference | 12 weeks
  Waist circumference as measured at midpoint between the lower rib and the iliac crest at the end of a normal expiration using a tap measure.
Lean Body Mass | 12 weeks
  Lean body mass (kg) was determined using a bioelectrical impedance-meter.
Glucose | 12 weeks
  Blood glucose concentrations were assessed with a glucose reagent kit.
Insulin | 12 weeks
  Serum insulin was evaluated using an enzyme-linked immunosorbent assay (ELISA) kit.
Homeostatic Model Assessment - Insulin Resistance | 12 weeks
  Homeostatic model assessment - insulin resistance was calculated from the fasting plasma blood glucose and insulin levels according to previously established models.

IPD SHARING:
Plan to Share IPD: No